CLINICAL TRIAL: NCT02498756
Title: A Study of Ipilimumab Plus Cytokine-induced Killer Immunotherapy for Stage II Melanoma Patients
Brief Title: Cytokine-induced Killer Study for Patients With Stage II Melanoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First People's Hospital of Changzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Melanoma001
Record Dates: First submitted 2015-06-30; First posted 2015-07-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IP plus CIK (Experimental): Patients receive ipilimumab and CIK.
  Interventions: Biological: Cytokine-induced killer cells; Drug: Ipilimumab
- IP alone (Active Comparator): Patients receive ipilimumab alone.
  Interventions: Drug: Ipilimumab

INTERVENTIONS:
Biological: Cytokine-induced killer cells — CIK cells are transferred every 3 months for 1 year.
  Arms: IP plus CIK
Drug: Ipilimumab — Ipilimumab are delivered every 3 weeks for one year

SUMMARY:
For investigators' current experimental clinical trial, patients are given 4 injections of ipilimumab, given 3 weeks apart x 4 injections with or without cytokine-induced killer therapy. Investigators propose to test this dual therapy in patients with melanoma who have known stage I, metastatic melanoma. Investigators hypothesize that this form of combinatorial immunotherapy will result in tumor stabilization or shrinkage, significant prolongation of progression-free, disease-free or overall survival compared to the use of ipilimumab alone

DETAILED DESCRIPTION:
despite the best clinical efforts and breakthroughs in biotechnology, most patients diagnosed with advanced stage melanoma continue to die from their disease. Reasons for this include: 1) patients are often diagnosed at a time when their melanoma has already spread to other sites such as the chest cavity, bone, liver, and brain limiting the options for surgical excision and 2) the cancer cells are resistant or become resistant to chemotherapy drugs used to treat the patient. Resistance to one type of chemotherapy agent often rapidly leads to resistance against many other chemotherapy drugs. These reasons are the major causes of cancer progression that are usually discussed when considering treatment options for patients with disease that continues to grow and spread. However, another important part of the body should be considered-- the immune system. Scientists have clearly shown that melanoma cells produce a number of abnormal proteins or abnormal amounts of certain proteins found in normal melanoma cells. Normally one would expect a patient to develop an immune response against these abnormal proteins found in their cancer and attack them much the way the investigators would fight off an infection from a foreign bacteria or virus. However, for reasons that scientists do not fully understand, the immune system fails to respond adequately to these abnormal proteins and does not destroy the melanoma cells. This human clinical trial proposes a new way to make the immune system recognize the cancer cells and encourages it to attack and destroy them.

In this project, the investigators have put a mouse gene into human melanoma cancer cells, so that those cells produce these abnormal sugar patterns and stimulate the immune system to attack the melanoma. This strategy works well to kill other human cancer cells in the laboratory, but it needs to be tried in melanoma patients to see if it will be effective and to determine if such a treatment causes any side effects. Investigators propose to test this new treatment in patients with melanoma to see if it can stop, slow or destroy tumors in these patients. Patients will be injected with an anti-tumor immunotherapy consisting of three types of dead human melanoma cancer cells that have been genetically altered to express the mouse gene responsible for making this abnormal sugar-protein on the cells.

In this Phase II Study, patients with early stage melanoma will undergo a series of intradermal injections with cytokine-induced killer therapy. These cell lines have been transduced with a recombinant. In addition to the cik therapy, some patients will also receive ipilimumab as an important component of this immunization strategy that will attempt to enhance and activate the host immune system to destroy growing tumor cells. Endpoints of the study include safety assessments, and clinical, tumor and immunological responses.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of melanoma. AJCC Stage IV (any T, any N, M1), metastatic, progressive, refractory, melanoma.

Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1. Serum albumin ≥3.0 gm/dL.

Exclusion Criteria:

* Age <18-years-old. Active CNS metastases or carcinomatous meningitis. Patients with CNS lesions that have been treated and who have no evidence of progression in the brain on CT/MRI for ≥1 month are eligible. Pregnant or nursing women due to the unknown effects of immunization on the developing fetus or newborn infant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-08; Primary Completion 2038-08 (Estimated); Study Completion 2040-08 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 5 years
Progression Free Survival (PFS) | 1 year